CLINICAL TRIAL: NCT04984941
Title: Evaluation of the Role of IgE Responses to Der p 1 and Der p 2 in Chinese House Dust Mite-Allergic Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-047
Record Dates: First submitted 2021-07-11; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Asthma; Allergic Rhinitis; Conjunctivitis; Atopic Dermatitis
Keywords: House dust mite; Der p 1; Der p 2; China
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Conjunctivitis; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One hundred patients were enrolled, based on sensitization and doctor-diagnosed allergy to HDM. Questionnaires were administered to document demographic and clinical characteristics. Serum IgE reactivity toDermatophagoides pteronyssinus (Dp) extract, Der p 1, Der p 2 and Der p 10 was measured by ImmunoCAP.

DETAILED DESCRIPTION:
Background: The role of specific IgE (sIgE) against Der p 1and Der p 2 in Chinese patients with house dust mite (HDM)allergy has not yet been well investigated.Methods: One hundred patients were enrolled, based on sensitization and doctor-diagnosed allergy to HDM. Questionnaires were administered to document demographic and clinical characteristics. Serum IgE reactivity toDermatophagoides pteronyssinus (Dp) extract, Der p 1, Der p 2 and Der p 10 was measured by ImmunoCAP.

ELIGIBILITY:
Inclusion Criteria:

* HDM-allergic patients reporting allergic rhinitis, conjunctivitis, asthma and/or atopic dermatitis and who had never undergone immunotherapy, were enrolled if they were sensitized to Dp as judged by ImmunoCAP ( ≥ 1 kU/l) and/or skin reaction index (SRI)by skin-prick test (SPT, a wheal diameter ≥ 0.5 mm).

Exclusion Criteria:

* Patients who refused to participate in the study.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All patients were evaluated by a physician face-to-face, using a detailed questionnaire to establish the nature and severity of their clinical manifestations. The questionnaire also included demographic characteristics, a family history of allergic diseases and any other history of allergic disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristics | 1 year
  Describe the patient's basic information in detail, including age, gender, family history, etc
Der p 1 Serum IgE | 1 year
  Prevalence of Der p 1 Serum IgE in HDM-Allergic Patients
Der p 2 Serum IgE | 1 year
  Prevalence of Der p 2 Serum IgE in HDM-Allergic Patients
Dp, Der p 1 and Der p 2 | 1 year
  Relationship between Serum IgE Levels of Dp, Der p 1 and Der p 2
Factors associated with specific IgE against Der p 1 | 1 year
  Study the patient's basic information and identify factors that are clearly associated with specific IgE against Der p 1
Factors associated with specific IgE against Der p 2 | 1 year
  Study the patient's basic information and identify factors that are clearly associated with specific IgE against Der p 2
the Number of Affected Organs | 1 year
  Association of Specific IgE Titers with the Number of Affected Organs

CONTACTS AND LOCATIONS:
Overall Officials: Wang Huiying, Study Chair — 2nd affiliated Hospital,School of Medicine,Zhejiang University,China
Locations (1):
- Second Affiliated Hospital，School of Medicine，Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No